CLINICAL TRIAL: NCT03155061
Title: Phase 1 Dose Escalating and Expansion Study of ONO-4578 Given as Monotherapy and Combinations of ONO-4578 and ONO-4538 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Study of ONO-4578 With and Without ONO-4538 in Subjects Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-01; jRCT2080223441 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2017-03-17; First posted 2017-05-16 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A (Dose Escalation Part): ONO-4578 monotherapy (Experimental): ONO-4578 specified dose on specified days in advanced or metastatic solid tumors
  Interventions: Drug: ONO-4578
- Part B: ONO-4578 in combination with ONO-4538 (Experimental): ONO-4578+ONO-4538 specified dose on specified days in advanced or metastatic solid tumors
  Interventions: Drug: ONO-4578; Drug: ONO-4538
- Part C (Expansion Part): ONO-4578 in combination with ONO-4538 (Experimental): ONO-4578+ONO-4538 specified dose on specified days in unresectable, advanced or recurrent gastric cancer
  Interventions: Drug: ONO-4578; Drug: ONO-4538
- Part D (Expansion Part): ONO-4578 in combination with ONO-4538 (Experimental): ONO-4578+ONO-4538 specified dose on specified days in unresectable, advanced or recurrent colorectal cancer
  Interventions: Drug: ONO-4578; Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4578 — ONO-4578 specified dose on specified days
Drug: ONO-4538 — ONO-4538 specified dose on specified days
  Arms: Part B: ONO-4578 in combination with ONO-4538; Part C (Expansion Part): ONO-4578 in combination with ONO-4538; Part D (Expansion Part): ONO-4578 in combination with ONO-4538

SUMMARY:
The objective of the study is to evaluate the safety, tolerability, pharmacokinetics, efficacy and biomarker of ONO-4578 and combinations of ONO-4578 and ONO-4538 in subjects with advanced or metastatic solid tumors and subjects with unresectable, advanced or recurrent gastric cancer, unresectable, advanced or recurrent colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumors (Part A, B)
* Unresectable, advanced or recurrent gastric cancer previously treated with anti-PD-(L)1 antibodies or naive to anti-PD-(L)1 antibodies (Part C)
* Unresectable, advanced or recurrent colorectal cancer(Part D)
* Life expectancy of at least 3 months
* Patients with ECOG performance status 0 or 1

Exclusion Criteria:

* Patients with severe complication
* Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety (adverse event, clinical laboratory test, 12-lead electrocardiography, chest X-ray, ECOG performance status) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Maximum observed serum concentration(Cmax) | Up to Cycle 1 (each cycle is 28 days)
Area Under the blood concentration-time Curve(AUC) | Up to Cycle 1 (each cycle is 28 days)
Half-life(T1/2) of ONO-4578 both alone and in combination with ONO-4538 | Up to Cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (22):
- Japan (22):
  - Aichi Clinical Site 1, Nagoya, Aichi-ken
  - Aichi Clinical Site 2, Toyoake, Aichi-ken
  - Chiba Clinical Site 1, Kashiwa, Chiba
  - Ehime Clinical Site1, Matsuyama, Ehime
  - Gunma Clinical Site 1, Ōta, Gunma
  - Hokkaido Clinical Site 1, Sapporo, Hokkaido
  - Iwate Clinical Site 1, Yahaba-cho, Iwate
  - Kanagawa Clinical Site 2, Sagamihara, Kanagawa
  - Kanagawa Clinical Site 1, Yokohama, Kanagawa
  - Osaka Clinical Site 2, Hirakata, Osaka
  - Osaka Clinical Site 3, Sakai, Osaka
  - Osaka Clinical Site 4, Takatsuki, Osaka
  - Saitama Clinical Site 2, Hidaka, Saitama
  - Saitama Clinical Site 1, Ina-machi, Saitama
  - Shizuoka Clinical Site 1, Nagaizumi-Cho, Shizuoka
  - Tokyo Clinical Site 1, Chuo-ku, Tokyo
  - Tokyo Clinical Site 4, Itabashi-ku, Tokyo
  - Tokyo Clinical Site 2, Koto-ku, Tokyo
  - Tokyo Clinical Site 3, Shinjyuku-ku, Tokyo
  - Fukuoka Clinical Site 1, Fukuoka
  - Fukuoka Clinical Site 2, Fukuoka
  - Osaka Clinical Site 1, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawazoe A, Yamaguchi K, Hamaguchi T, Narita Y, Boku S, Oshima T, Hara H, Hamamoto Y, Ishido K, Esaki T, Hosaka H, Yasui H, Koeda K, Nishina T, Tsuji Y, Fukagawa T, Goto M, Oki E, Sugimoto N, Matsuoka H, Yokoyama F, Yoshida T, Yoshida K, Oshima Y, Iwasa S. ONO-4578 Plus Nivolumab in Unresectable Advanced or Recurrent Gastric or Gastroesophageal Junction Cancer. Cancer Sci. 2025 Sep;116(9):2523-2536. doi: 10.1111/cas.70130. Epub 2025 Jul 6. PMID 40618725
- [Derived] Iwasa S, Koyama T, Nishino M, Kondo S, Sudo K, Yonemori K, Yoshida T, Tamura K, Shimizu T, Fujiwara Y, Kitano S, Shimomura A, Sato J, Yokoyama F, Iida H, Kondo M, Yamamoto N. First-in-human study of ONO-4578, an antagonist of prostaglandin E2 receptor 4, alone and with nivolumab in solid tumors. Cancer Sci. 2023 Jan;114(1):211-220. doi: 10.1111/cas.15574. Epub 2022 Nov 4. PMID 36082616